CLINICAL TRIAL: NCT07125391
Title: Chemotherapy Combined With Propranolol Hydrochloride as Neoadjuvant Therapy for Advanced High-grade Serous Ovarian Cancer: A Prospective, Multicenter, Phase II Clinical Study
Brief Title: Chemotherapy Combined With Propranolol Hydrochloride as Neoadjuvant Therapy for Advanced High-grade Serous Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bai-Rong Xia (Other)
Responsible Party: Sponsor-Investigator, Bai-Rong Xia, Chairman of Department of Gynaecology Surgery, Anhui Provincial Cancer Hospital
Organization: Anhui Provincial Cancer Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LLYJ-0015
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
Keywords: NACT
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects who met the inclusion and exclusion criteria were divided into 2 groups:
  Cohort A received propranolol hydrochloride (20mg, BID, QD), paclitaxel/paclitaxel liposome (135-175mg/m2, d1, Q3W), carboplatin (AUC=4-5, d1, Q3W) for 3-4 cycles of neoadjuvant therapy. Subsequently, interval debulking surgery (IDS) was performed. Propranolol hydrochloride was taken one week before neoadjuvant therapy.
  Cohort B received neoadjuvant paclitaxel/paclitaxel liposome (135-175mg/m2, d1, Q3W) and carboplatin (AUC=4-5, d1, Q3W) for 3-4 cycles, followed by interval debulking surgery (IDS).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): Received paclitaxel/paclitaxel liposome (135 - 175mg/m2, d1, Q3W), carboplatin (AUC=4-5, d1, Q3W), neoadjuvant therapy for 3 - 4 cycles, followed by interval debulking surgery (IDS)
  Interventions: Drug: Cohort A

INTERVENTIONS:
Drug: Cohort A — received propranolol hydrochloride (20mg, BID, QD), paclitaxel/paclitaxel liposome (135-175mg/m2, d1, Q3W), carboplatin (AUC=4-5, d1, Q3W) for 3-4 cycles of neoadjuvant therapy. Subsequently, interval debulking surgery (IDS) was performed. Propranolol hydrochloride was taken one week before neoadjuvant therapy

SUMMARY:
Ovarian Cancer (OC) is one of the most common gynecological malignant tumors. In recent years, the incidence of ovarian cancer in China has been on the rise, but its mortality ranks the first among gynecological tumors. Cytoreductive Surgery (CRS) combined with chemotherapy is the standard treatment for patients with advanced ovarian cancer. However, most of the ovarian cancer is stage Ⅲ and above, and there may be a certain degree of organ metastasis. Preclinical studies have found that the stress of melanoma block beta adrenergic signals in mice, which USES beta blockers, checkpoint will enhance resistance to PD - 1 the activity of the inhibitor, to improve the treatment of mice on the immune response. Non-selective β-blockers can also improve the efficacy of melanoma immunotherapy. Retrospective studies have shown that incidental use of β-blockers in combination with antiangiogenic agents, chemotherapy, and immune therapy can prolong DFS, PFS, and OS in cancer patients. A large, multicenter retrospective study found that ovarian cancer patients who took nonselective β-blockers for hypertension had better survival than those who did not. In conclusion, this study aims to explore new auxiliary chemotherapy combined propranolol treatment of high efficacy and safety of ovarian cancer, provide more evidence-based basis for clinic.

DETAILED DESCRIPTION:
The study included patients with inoperable stage III or IV ovarian cancer who were initially treated in FIGO stage III or IV. "A phase II trial to explore the efficacy and safety of neoadjuvant chemotherapy plus propranolol in patients with histologically confirmed high-grade serous ovarian cancer." Na row standard subjects were divided into 2 groups: Queue A accept propranolol hydrochloride (20 mg, BID, QD), paclitaxel/paclitaxel liposome (135-175 mg/m2, d1, Q3W) and carboplatin (AUC = 4-5, d1, Q3W), neoadjuvant therapy cycle, A total of 3-4 Subsequently, interval debulking surgery (IDS) was performed. Propranolol hydrochloride was taken one week before neoadjuvant therapy. Queue B receive paclitaxel/paclitaxel liposome (135-175 mg/m2, d1, Q3W) and carboplatin (AUC = 4-5, d1, Q3W), neoadjuvant therapy cycle, a total of 3-4 line then intermittent tumor cells to destroy the loss (interval debulking surgery, IDS); Patients will accept the tumor assessment before the surgery, postoperative by researchers according to aid in the treatment of ovarian cancer guidelines take corresponding.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was obtained before any trial-related procedures were performed.
* Women, 18 to 75 years old;
* FIGO stage for stage III or IV, including not surgery in patients with stage III or IV beginning for ovarian cancer; Histopathology confirmed high-grade serous ovarian cancer.
* According to the response evaluation criteria in 1.1 (RECIST1.1) definition, patients must have a measurable lesions
* Agreed to provide the participants formalin fixed and tumor tissue specimens or fresh biopsy tissue tumor lesions markers detection
* ECOG score 0-1 points
* Expected survival time 6 months or more
* Enough organ function, without severe hematopoietic dysfunction and heart, lung, liver, kidney dysfunction, and immune deficiency, participants need to satisfy the following laboratory indicators

  * hemoglobin (HGB) 90 g/L or higher
  * Neutrophils (NEUT) acuity 1.5 x 109 / L or white blood cell count (WBC) or 3 x 109 / L
  * Platelet (PLT) or 90 x 109 / L
  * Nmda aminotransferase (AST) 2.5 x ULN or less
  * Alanine aminotransferase (ALT) 2.5 x ULN or less
  * Total bilirubin (TBIL) 1.5 x ULN or less
  * Serum creatinine (SCr) 1.0 x ULN or less
  * Potential fertility women in the group of 7 days before the serum or urine HCG were negative (postmenopausal women considered must be at least 12 months of amenorrhea fertility; Pregnancy tests are not required for women with documented tubal ligation)
  * Potential fertility women are willing to take in the experiment of the medical contraception

Exclusion Criteria:

* Malignant diseases other than ovarian cancer (excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, and/or radical resection in situ carcinoma) diagnosed within 5 years before the first dose
* Current are participating in clinical research and treatment of intrusive, or within 4 weeks before the first dose received study used drugs or other treatments
* Always received pelvic radiotherapy and systemic chemotherapy for ovarian cancer, tumor targeting therapy, immune therapy
* Need treatment of symptomatic or non-control brain metastasis at the same time, including but not limited to, surgery, radiation and/or corticosteroids, or with the clinical manifestations of spinal cord compression
* Current use of oral or intravenous beta blockers (atenolol, peso parlour, carvedilol and labetalol, metoprolol, than the parlour, his law such as beta blockers) cannot safely use of propranolol
* Patients with contraindications to β-blockers were excluded according to the contraindications in the propranolol package insert.
* Patients were receiving systemic glucocorticoids (excluding topical glucocorticoids by nasal spray, inhalation, or other route) or any other form of immunosuppressive therapy within 7 days before the first study dose; Note: allows the use of physiological doses of corticosteroids (10 mg/day or less prednisone or equivalent drugs)
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
* Patients who were allergic to the active ingredient or excipients of propranolol hydrochloride in this study
* Have not fully recovered from any intervention-related toxicity and/or complications before starting treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or alopecia)
* Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive)
* Hepatitis b patients with known
* Activity of HCV infection subjects (HCV antibody positive and HCV - RNA levels higher than the detection limit)
* For the first time to give medicine before (1 cycle, day 1) vaccinated live vaccine within 30 days
* Pregnant or lactating women
* Any serious or uncontrolled systemic disease, such as

  * resting electrocardiogram (ecg) in rhythm, conduction, or have a significant and severe symptoms to appear on the form is hard to control the exceptions, such as complete left bundle branch block, Ⅱ degrees above heart block, ventricular arrhythmia or atrial fibrillation
  * Unstable angina and congestive heart failure, New York heart association (NYHA) classification of grade 2 or more chronic heart failure
  * Within 6 months before the selected treatment had any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, etc.
  * First dose exist within 1 year before need to glucocorticoid treatment of infectious pneumonia history, or the current clinical activity interstitial lung disease; Active tuberculosis
  * There need systemic treatment of active or failure to control the infection
  * Clinical activity diverticulitis, abdominal abscess, gastrointestinal obstruction
  * Liver disease such as cirrhosis of the liver, decompensated liver disease, acute or chronic active hepatitis
  * Mental disorders and unable to cooperate with treatment
* Any medical history or evidence of illness, abnormal treatment or laboratory values, or other conditions that might interfere with the results of the trial or prevent full participation in the study, or any other potential risk that might be considered by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
CRS | 3-month
  Chemotherapy Response Scoring：Pathological assessment was conducted on the retinal tissue removed during the surgery

SECONDARY OUTCOMES:
R0 resection rate | 3-month
  the percentage of patients received R0 resection after neoadjuvant therapy
Overall Response Rate (ORR) After Neoadjuvant treatment | 3-month
  Overall Response Rate according to RECIST1.1 after Neoadjuvant treatment. ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions
Pathological complete remission rate | 3-month
  No residual invasive carcinoma was found under the microscope, but ductal carcinoma in situ could be found; In addition, compare the amount of cancer cells in the specimen before and after the new adjuvant therapy, and use of the Miller Payne grading system to evaluate the effect of the new adjuvant therapy
12-month disease-free survival rate | 12 months
  The rate of patients who did not have any event from the beginning of enrollment to 12 months, including disease progression, inoperable, local or remote recurrence, and death from any cause
12-month survival rate | 12 months
  Rate of patients who did not have a death event from enrollment to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Rong Xia, Doctor, Study Chair — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui Cancer Hospitail, Hefei, Anhui, China